CLINICAL TRIAL: NCT06279754
Title: Recombinant Human Endostatin Combined With Evafolimab Injection and Synchronal Radiochemotherapy for First-line Treatment of Locally Advanced Stage III Squamous Non-small Cell Lung Cancer
Brief Title: Recombinant Human Endostatin Combined With Envafolimab and Synchronal Radiochemotherapy
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZLXGBXKYXM-031-01
Record Dates: First submitted 2024-01-29; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Locally Advanced Squamous Non-small Cell Lung Cancer
Keywords: recombinant human endostatin; envafolimab; synchronal radiochemotherapy
MeSH Terms: interventions — Endostatins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- recombinant human endostatin Group (Experimental): Recombinant human endostatin and enrolizumab injection combined with Synchronal Radiochemotherapy
  Interventions: Drug: Recombinant Human Endostatin Injection

INTERVENTIONS:
Drug: Recombinant Human Endostatin Injection — Recombinant Human Endostatin Injection：210 mg, intravenous infusion for 72 hours, once every three weeks cycle Evafolimab Injection：Subcutaneous injection on day 1, 8, and 15, once every three weeks cycle
  Other Names: Evafolimab Injection

SUMMARY:
This study is a prospective, single arm, single center open clinical study aimed at evaluating the efficacy and safety of recombinant human endostatin and envafolimab combined with synchronal radiochemotherapy in patients with locally advanced squamous non-small cell lung cancer who cannot undergo surgery in stage III.

DETAILED DESCRIPTION:
This study is a prospective, single arm, single center open clinical study aimed at evaluating the efficacy and safety of recombinant human endostatin and envafolimab combined with synchronal radiochemotherapy in patients with locally advanced squamous non-small cell lung cancer who cannot undergo surgery in stage III.

Patients with locally advanced stage III squamous non-small cell lung cancer who have not received systematic treatment in the past and cannot be treated surgically, after signing informed consent, qualified subjects who meet the inclusion criteria will be screened. They will receive 2 cycles of recombinant human endostatin combined with envafolimab and platinum containing chemotherapy. Radiotherapy will be carried out simultaneously in cycles 1-2, and after 2 cycles, they will receive maintenance treatment with envafolimab until the disease progresses and intolerable toxicity is detected, The treatment period does not exceed 12 months

ELIGIBILITY:
Inclusion Criteria:

* The patient voluntarily participated in this study, voluntarily underwent treatment and follow-up, and signed an informed consent form;
* According to the International Association for the Study of Lung Cancer and the Joint Committee on Cancer Classification, 8th edition of the TNM staging classification for lung cancer, locally advanced and unresectable stage III non-small cell lung cancer with histopathological diagnosis;
* According to the criteria for evaluating the efficacy of solid tumors (RECIST 1.1), there should be at least one imaging measurable lesion; Patients who have not received PD-1/PD-L1 antibody treatment in the past.
* 18-70 years old; ECOG PS score: 0-1 points; Expected survival period exceeding 3 months;
* Main organ functions meet treatment standards
* Women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives, or condoms) during the study period and within 6 months after the end of the study; Within 7 days prior to enrollment in the study, the serum or urine pregnancy test was negative and must be a non lactating patient; Men should agree to patients who must use contraceptive measures during the study period and within 6 months after the end of the study period.

Exclusion Criteria:

* Patients who have previously received PD-1/PD-L1 antibody treatment;
* Respiratory syndrome caused by pleural effusion or ascites (according to NCICTCAE classification ≥ grade 2 dyspnea;
* Patients with brain metastases accompanied by symptoms or symptom control time less than 2 months;
* Has experienced or currently suffers from other malignant tumors within 5 years;
* Within the first 4 weeks of grouping or during the medication period of this study, it is planned to undergo systemic anti-tumor therapy, including cytotoxic therapy and targeted drug therapy. Received radiotherapy within 4 weeks prior to grouping;
* Patients with any severe and/or uncontrolled diseases
* Received significant surgical treatment, open biopsy, or obvious traumatic injury within 28 days prior to grouping;
* Patients with any signs of bleeding or medical history, regardless of severity; Within the first 4 weeks of grouping, patients with any bleeding or bleeding events ≥ CTCAE level 3, with unhealed wounds, ulcers, or fractures;
* Individuals who have experienced arterial/venous thrombosis events within 6 months, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis, and pulmonary embolism;
* Individuals with a history of psychiatric drug abuse who are unable to quit or have mental disorders;
* Participated in clinical trials of other anti-tumor drugs within four weeks;
* According to the researcher's judgment, there are accompanying diseases that seriously endanger patient safety or affect patient completion of the study;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-18 (Estimated); Primary Completion 2024-06-18 (Estimated); Study Completion 2025-12-18 (Estimated)

PRIMARY OUTCOMES:
objective response rate | After 6 weeks
  After treatment, the ratio of patients assessed as CR and PR according to RECIST 1.1

SECONDARY OUTCOMES:
Overall survival | The time from the start of treatment to death or last follow-up
  The time from the start of treatment to death or last follow-up
Progression-free survival | The time from the start of treatment to the first recording of disease progression
  The time from the start of treatment to the first recording of disease progression.

IPD SHARING:
Plan to Share IPD: Yes
Share mid-term data results and final data analysis results
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Half a year to one year after the start of the research
Access Criteria: All can be accessed